CLINICAL TRIAL: NCT07379515
Title: Effects of Topical Anesthesia Approaches on Dental Pain During and After Restorative Management of Dental Caries - Randomized Clinical Trial
Brief Title: Effects of Topical Anesthesia Approaches on Dental Pain During and After Restorative Management of Dental Caries
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dubai Health (Other Government)
Responsible Party: Principal Investigator, Sameeha Husain Al Marzooqi, Consultant, Dubai Health
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MBRU IRB-2024-695
Record Dates: First submitted 2025-12-08; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2025-12

CONDITIONS: Pulpitis; Pain Management
MeSH Terms: conditions — Pulpitis; Agnosia | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Non-medicated anelgesia (Experimental)
  Interventions: Device: Photobiomodulation (PBM)-induced analgesia device using multi-wavelength LED
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo
- Medicated anelgesia (Active Comparator)
  Interventions: Other: Medicated analgesia

INTERVENTIONS:
Device: Photobiomodulation (PBM)-induced analgesia device using multi-wavelength LED — Photobiomodulation (PBM)-induced analgesia device using multi-wavelength LED
  Arms: Non-medicated anelgesia
Other: Medicated analgesia — Topical anesthesia (Benzocaine 20%)
  Arms: Medicated anelgesia
Other: Placebo — Placebo with no intervention.
  Arms: Placebo

SUMMARY:
The purpose of the Research Study and Overview of Participation: This study will compare different approaches used to prevent pain when giving local anesthesia to numb the teeth while managing dental cavities and decay. Specifically, it seeks to determine which approach will reduce the pain and discomfort during or after the procedure. This will help dentists to choose the best approach to reduce patient's pain and discomfort and improve the overall experience of dental treatment.

Participants in the study would likely undergo the following:

1. Screening and Consent: Participants would be assessed for eligibility (e.g., age, health status, and presence of dental caries requiring treatment) and would provide informed consent.
2. Intervention: Participants would be randomly assigned to different groups based on the type or method of topical anesthesia being tested.
3. Treatment Procedure: Dental caries management would be performed under local anesthesia, with the designated topical anesthetic applied beforehand.
4. Pain Assessment: Participants would rate their pain levels during and after the procedure using validated pain measurement scales (e.g., visual analog scale).
5. Follow-Up: Participants might be monitored for a short duration post-treatment to assess any residual pain or side effects.

This design ensures that the study collects reliable data on the effectiveness of the different topical anesthetic approaches while prioritizing patient safety and comfort.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants: American Society of Anesthesiology Class I or II
* Adults aged 18-59 years
* No history of allergy to local anesthesia or excipients included in the vial
* Participant requiring caries management for a maxillary premolar tooth (ICDAS I-V), with reversible pulpitis.

Exclusion Criteria:

* American Society of Anesthesiology Class III or higher
* Participants with systemic conditions affecting pain perception
* Participants on chronic pain medication
* Pregnant or breastfeeding women
* History of allergy to topical/local anesthesia
* Taking any analgesic 48 hours before testing, such as an NSAID, opioids, or
* acetaminophen
* Recent oral trauma
* Deep carious lesion with irreversible pulpitis or pulpal necrosis

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 204 (Estimated)
Dates: Start 2026-01-02 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Pain score after local anesthesia administration, dental procedure, and 48 hours postoperatively. | Within 5 minutes after local anesthesia administration, during dental procedure, directly after finishing the procedure, and 48 hours postoperatively.
  Pain score based on Visual Analog Scale (1-10) with highest score indicates the most severe pain.

SECONDARY OUTCOMES:
Pain score with prick pain test (PPT) | One minute after topical anesthesia.
  Pain score will be reported as "pain" or "no pain".
Pain score with pulpal stimulation using electric pulp tester (EPT) | After 2 minutes of topical anesthesia.
  Digital reading from 1 to 64 with the highest score indicates no pain response on electric stimulation.
Amount of local anesthesia to be given | At the end of dental procedure.
  Counting the number of used local anesthetic carpules.
Need for additional analgesics | Within 48 hours postoperatively.
  Count the number and dose of oral analgesics taken by the patient.
Reporting of any adverse effects, such as mucosal irritation, allergic reactions, and delayed pain relief. | Within 48 hours postoperatively.
  Reported by the patient.

IPD SHARING:
Plan to Share IPD: No